CLINICAL TRIAL: NCT00002079
Title: Phase II Study of the Safety and Surrogate Marker Efficacy of Butyldeoxynojirimycin (SC-48334) and AZT in Symptomatic HIV-1 Infected Patients With 200 - 500 CD4+ Cells/mm3. (NOTE: Asymptomatic HIV-1 Infected Patients Also Eligible)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: G D Searle (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 057B; NS8-91-02-009
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1993-03

CONDITIONS: HIV Infections
Keywords: Zidovudine; 1-Deoxynojirimycin
MeSH Terms: conditions — HIV Infections | interventions — miglustat; Zidovudine

INTERVENTIONS:
Drug: Butyldeoxynojirimycin
Drug: Zidovudine

SUMMARY:
To assess the dose-related antiviral effects of SC-48334 and zidovudine (AZT) administered in combination or individually in HIV-1 positive patients with 200 - 500 CD4+ cells/mm3. To determine the safety of escalating doses of SC-48334 when administered in combination with any of three doses of AZT to symptomatic HIV-1 positive patients with 200 - 500 CD4+ cells/mm3, and to assess the pharmacokinetics of the two drugs, given separately and in combination.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Documented HIV infection.
* CD4 cell count 200 - 500 cells/mm3.
* Prior therapy with 12 - 48 weeks of AZT.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Clinically significant diarrhea without definable cause (> 3 liquid stools per day for more than 7 days within 6 months prior to study entry).
* Diarrhea, as above, with known non-HIV-related cause occurring within 1 month prior to study entry.
* Symptoms meeting CDC criteria for AIDS classification.
* Fever as a constitutional sign of HIV disease (> 38.5 degrees C persisting for more than 14 consecutive days or for more than 15 days in any given 30-day period prior to study entry).
* Malignancies, other than basal cell carcinoma and Kaposi's sarcoma (provided patient has fewer than 10 Kaposi's sarcoma lesions, no non-skin lesions, and no requirement for systemic treatment).
* Significant organ dysfunction.
* Known hypersensitivity to SC-48334 or AZT or related compounds.

Concurrent Medication:

Excluded:

* Any investigational drug other than SC-48334.
* Any anti-HIV drug other than AZT.
* Cancer chemotherapy.

Patients with the following prior conditions are excluded:

* History of cataracts or known increased risk of cataract formation.
* Known hypersensitivity to SC-48334 or AZT or related compounds.
* History of lactose intolerance.

Prior Medication:

Excluded:

* Prior SC-48334.
* Cancer chemotherapy within 6 months prior to study entry.
* Treatment with any investigational drug or any drug with anti-HIV activity, other than AZT, within 30 days prior to study entry.

Prior Treatment:

Excluded:

Whole-body irradiation within 6 months prior to study entry. Current use of illicit substances, or abuse of alcohol, which would limit compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Dr Marcus Conant, San Francisco, California
  - Shared Med Research Foundation, Tarzana, California
  - Stratogen of South Florida, Miami Beach, Florida
  - Saint Joseph's Hosp / Infectious Disease Rsch Institute, Tampa, Florida
  - West Paces Clinical Research Incoporated, Atlanta, Georgia
  - Dr Samuel W Golden, Pittsburgh, Pennsylvania
  - Dallas Veterans Administration Med Ctr, Dallas, Texas
  - Dr Daniel Barbero, Fort Worth, Texas
  - Park Plaza Hosp, Houston, Texas

REFERENCES:
- [Background] Fischl MA, Resnick L, Coombs R, Kremer AB, Pottage JC Jr, Fass RJ, Fife KH, Powderly WG, Collier AC, Aspinall RL, et al. The safety and efficacy of combination N-butyl-deoxynojirimycin (SC-48334) and zidovudine in patients with HIV-1 infection and 200-500 CD4 cells/mm3. J Acquir Immune Defic Syndr (1988). 1994 Feb;7(2):139-47. PMID 7905523